CLINICAL TRIAL: NCT06015594
Title: Metformin Treatment in Adolescent Patients With PCOS: A Long-term, Winning Metabolic Choice. Results From a Single Center 5-years Retrospective Clinical Study
Brief Title: Metformin Treatment in Adolescent Patients With PCOS: A Long-term, Winning Metabolic Choice.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Di Michele, Principal investigator (Medical doctor), University of Cagliari
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PG/2020/12426
Record Dates: First submitted 2023-08-03; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: insulin resistance; metformin; adolescents
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin group (Experimental): Treated with metformin
  Interventions: Drug: Metformin
- Control group (No Intervention): not treated

INTERVENTIONS:
Drug: Metformin — Patients treated with metformin
  Arms: Metformin group

SUMMARY:
This study aimed to understand whether metformin therapy can improve insulin resistance in adolescent PCOS patients, both during treatment and after discontinuation, and to evaluate its action on the hormonal and metabolic pathways.

DETAILED DESCRIPTION:
Data were retrospectively retrieved from a database of clinical data collected in the Outpatient Pediatric and Adolescent Gynecology Clinic of the University Hospital "Duilio Casula," Monserrato, Cagliari (Division of Gynecology and Obstetrics, Department of Surgical Sciences, University of Cagliari, Italy), between 2015 and 2019. PCOS diagnosis was adapted for age following the 2019 update from Witchel SF and Carmina's recommendation.

The population consisted of 168 PCOS patients aged 12 to 17. Clinical examination, medical history, blood sampling, and pelvic ultrasound (US) were performed. The number of post-menarche years and the body mass index (BMI) were collected.

The patients were subjected to physical examination to evaluate hirsutism, according to the criteria of the Ferriman and Gallwey score, as well as acne, using the Cremoncini classification.

Each participant received detailed advice on improving their lifestyle, such as physical activity and nutrition. Investigators gave indications of the various food and their weighted intake and a balanced composition of macronutrients (carbohydrates 55%, lipids 25%, protein 20%; fiber ≥25 g/day), as recommended by the Reference intake levels of nutrients and energy for the Italian population (LARN) guidelines. Vegetables, fruit, cereals, fish, and pulses, typical of the Mediterranean style, were included in the diet.

Investigators recommended ≥150 minutes per week of moderate or ≥75 minutes of vigorous-intensity exercise for weight gain prevention, minimizing sedentary time, and including strength training exercises for two days per week, as reported from the 2018 PCOS guideline.

Laboratory evaluations were performed during the menstrual cycle's first follicular phase (days 3-7) and after a fast of 10-12 hours. Menstrual bleeding was induced by administering medroxyprogesterone acetate (10 mg/day for five days) in amenorrhoeic patients.

Follicle-stimulating hormone (FSH), luteinizing hormone (LH), 17-β estradiol (E2), total testosterone (TT), delta-4-androstenedione (A), 17-hydroxyprogesterone (17-OH-P) and sex hormone binding globulin (SHBG) were tested. In addition, total cholesterol, HDL, LDL, and triglycerides were measured with these blood tests.

The following day, the patients underwent a 75 g oral glucose tolerance test (OGTT). The OGTT was performed at 9 am after fasting overnight. Blood samples were collected basally and 60, 90, 120, and 180 min after ingesting 75 g of glucose in 150 ml of water. Insulin and glucose were assayed in all samples. Serum E2, FSH, LH, and TT were measured by chemiluminescence immunoassay Immulite (Siemens Products Corporation, Los Angeles, CA). Enzymatic methods were used for glucose, cholesterol, and triglycerides determination. Radioimmunoassay (RIA) was used to measure serum A, insulin and 17-OHP (Diagnostic System Laboratories, Inc. [DSL], Webster, TX). Insulin and glucose values were expressed as the area under the curve (AUC). The AUC was calculated using the trapezoidal rule method and reported as mIU/ml times 180 min for insulin.

A normal glycemic response to OGTT was defined according to the criteria of the National Diabetes Data Group (1979).

As previously described, a normal insulinemic response to OGTT was defined by a threshold AUC value of 16,900 mIU / ml / 180 min.

Insulin sensitivity evaluation was estimated using the homeostatic model assessment index (HOMA), which was calculated as follows: HOMA = [fasting insulin (mU/ml) * fasting glucose (mmol/l)/22, 5].

The same operator acquired ovarian morphology and ovarian volume for all patients. Ultrasound was performed by a transabdominal probe in a whole bladder or transvaginally. A Voluson E6 ultrasound system equipped with a 2-8 MHz RAB4-8-D convex transducer (GE Medical Systems, Austria) was used for the investigation. The ultrasound examination was performed on the same day the blood samples were taken. Ovarian volume was calculated using the formula for a modified prolate ellipsoid (longitudinal x transverse x anterior-posterior * 0.5233). The mean volume values of both ovaries were included in the statistical analysis.

Participants were categorized into two groups: the study group, consisting of patients who received metformin therapy, and the control group, which did not receive metformin during the study period.

The metformin dose was determined based on the study by Fulghesu et al. Both the study and control group underwent the same combined oral contraceptive pills (COCs), containing drospirenone 3 mg/ethinyl estradiol 20 μg (3 mg DRSP/20 μg EE-24/4).

Follow-up was performed every 3-6 months in the first year, then after 12 months by OGTT and clinical evaluation.

After about 24 months of treatment, the patients returned to the hospital and repeated clinical and laboratory examinations. Finally, the patients repeated the same blood tests and overall assessment at least 24 months after discontinuing metformin therapy. Baseline data are expressed as b-AUC, b-HOMA, and b-BMI. End-of-therapy evaluation data are described as e-AUC, e-HOMA, and e-BMI.

Evaluation data after the end of therapy are reported as ae-AUC, ae-HOMA, and ae-BMI.

Patient data were collected anonymously on an Excel® database (Office 365). Statistical analysis was performed using the IBM SPSS Statistics statistical software, version 26 (IBM SPSS Statistics, Chicago, IL, USA). Measurement data corresponding to the normal distribution were expressed by mean ± SD, and the t-test was used for the paired samples (Student's t-test). In addition, the count data were expressed as n (%), and the beta coefficient of linear regression with a 95% confidence interval (95% CI) was reported for each analysis. In all calculations, a p-value < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria: Pcos Adolescents

-

Exclusion Criteria:

Other type of hyperandrogenism

Ages: 10 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Insulin resistance change in eighty hyperinsulinemic patients after metformin therapy and its discontinuation | about 3 years
  To verify metformin treatment's immediate and long-term efficacy in hyperinsulinemic adolescent patients with PCOS and the evolution of metabolic status after treatment discontinuation.
Androgen levels change in eighty hyperinsulinemic patients after metformin therapy and its discontinuation | about 3 years
  To compare changes in androgen plasmatic levels such as total testosterone (TT) and delta-4-androstenedione (A) between the hyperinsulinemic adolescent patients with PCOS and the control group who have not received the metformin treatment by immediate and secondary assessment at the end of treatment of androgen plasmatic levels.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-07-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT06015594/Prot_SAP_ICF_000.pdf